CLINICAL TRIAL: NCT02876549
Title: G6PD Assessment Before Primaquine for Radical Treatment of Vivax Malaria
Acronym: GAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Nangarhar University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BAKMAL1601
Record Dates: First submitted 2016-07-28; First posted 2016-08-23 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Vivax Malaria
Keywords: G6PD; Primaquine
MeSH Terms: conditions — Malaria, Vivax | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G6PD Normal (Experimental)
  Interventions: Drug: Chloroquine; Drug: Primaquine 0.25 mg/kg/day
- G6PD Deficient (Experimental)
  Interventions: Drug: Chloroquine; Drug: Primaquine 0.75 mg/kg weekly

INTERVENTIONS:
Drug: Chloroquine — 10 mg/kg on day 0 & 1 and 5mg/kg on day 2, (Afghanistan NMLCP guidelines)
Drug: Primaquine 0.25 mg/kg/day — 0.25 mg/kg/day for 14 days
  Arms: G6PD Normal
Drug: Primaquine 0.75 mg/kg weekly — 0.75 mg/kg weekly for eight weeks
  Arms: G6PD Deficient

SUMMARY:
This will be a single-arm observational cohort study. Malaria patients with Plasmodium vivax and meeting study inclusion criteria, who give consent to be enrolled in the study, will have their G6PD status measured by the CareStart™ G6DP rapid diagnostic test (G6PD RDT), and primaquine prescribed according to the result. According to the G6PD RDT result, primaquine will be prescribed at 0.25mg/kg/day for 14 days (normal patients) or 0.75mg/kg weekly for eight weeks (deficient patients). All will receive treatment with chloroquine to clear asexual stages of infection.

Patients will be reviewed at day 2, day 7 and day 14. At these visits patients will undergo a brief clinical assessment and a small blood sample will be taken for repeat haemoglobin measurement and dried blood spot for carboxyprimaquine measurement (day 7 and day 14 only).

In general, antimalarial treatment will be unsupervised to reflect field conditions. However a subset of 25 G6PD normal patients at a single site will have each day of their primaquine treatment administered and observed at the treatment centre. This is to determine a calibration curve for primaquine pharmacokinetic studies.

Dried blood spots will be stored appropriately. Day zero samples will be genotyped in Bangkok (MORU, Dr. Mallika Imwong) after DNA extraction. PCR-RFLP will be used to detect the allele associated with the Mediterranean variant of G6PD deficiency. In addition DNA extracts will be sent for more systematic genetic testing for known G6PD variants through existing collaborations with the Wellcome Trust Sanger Institute. The day 7 and 14 dried blood spot samples will be analysed in the MORU pharmacology laboratory for primaquine and carboxyprimaquine concentrations, from which adherence to primaquine can be determined retrospectively, using the subset of 25 patients receiving directly observed therapy to calibrate the results.

Funder: WellcomeTrust, Grant reference: 107548/Z/15/Z

DETAILED DESCRIPTION:
1. Screening All patients registering for outpatient services in the outpatient department will undergo routine investigation. When malaria is suspected, a thick and thin blood smear will be obtained for microscopic diagnosis of Plasmodium vivax or a malaria RDT undertaken. After the diagnosis is confirmed microscopically, an assessment will be made to see if the patient fulfils the study inclusion and exclusion criteria.

   The following clinical screening procedures will be performed. The age, gender, ethnic group, and contact details of the subject will be recorded in the source documents. In the medical history, any history of chronic disease including previous history of haemolysis or anaemia will be noted along with a history of allergy to any medications (including chloroquine or primaquine).

   Pregnancy is a contraindication to primaquine and all women considered at risk of pregnancy will undergo urine pregnancy testing prior to enrolment. A pregnancy test is done routinely in Afghanistan, consistent with National Treatment Guidelines.

   Vital signs (axillary temperature in degrees Celsius, heart rate, respiratory rate, blood pressure, and weight in kilograms) will be recorded. The physician will perform a general systems examination.
2. Consent Patients who fulfil the study inclusion and exclusion criteria will be approached for informed consent.
3. Procedures after enrolment

   Once informed consent is given, a second capillary blood sample (finger prick) will be taken for:
   * CareStart RDT G6PD test. The RDT will be read at the appropriate time (10 minutes) and the result noted in the source documents. The RDT itself will be labelled and retained for future reference. It can also be analysed for host and parasite genotypes.
   * Baseline haemoglobin measurement via the HemoCue system. This will generally involve use of a micropipette and the HemoCue microcuvettes.
   * Collection of a dried blood spot (FTA card) labelled with an individual barcode.
   * If a malaria RDT was used for diagnosis this will also be labelled and kept if possible for future analyses of G6PD and parasite genotyping.
   * Biosensor recordings will also be made in a subset of patients at day 0 and day 14, if and when the device becomes available. These results will not influence patient management which will be based only on the RDT result.
4. Antimalarials Chloroquine will be provided aiming for a dose of 10 mg/kg on day 0 & 1 and 5mg/kg on day 2, (Afghanistan NMLCP guidelines).

   Primaquine will also be provided. (See dosing tables below) The target dose of primaquine is:
   * 0.25 mg/kg/day for 14 days (G6PD normal patients)
   * 0.75 mg/kg weekly for eight weeks (G6PD deficient patients). For small children, accurate drug dosage will be ensured by crushing a whole 15mg tablet and mixing in 10 ml water (with sugar if possible) prior to oral administration of 1-4 ml via a syringe (see Table 2). For older children and smaller adults tablets will be split to the nearest quarter (see Appendix these doses can also be crushed for administration if necessary).

   Primaquine daily dosing This dosing table provides a daily dose of between 0.19 and 0.33 mg/kg primaquine (total dose over 14 days 2.6 - 4.7 mg/kg).

   Children will be offered sweet drinks once the drug been administered to minimize the chance of vomiting. Parents of children will be shown how to measure the dose to allow accurate home administration.

   Treatment will generally be unsupervised to reflect field conditions. Sufficient primaquine will be given to last until the next visit. From the investigators own work and that of others in a similar population, adherence in this population is good, but this will be checked by pharmacological assessments of carboxyprimaquine levels.

   A subset of 25 G6PD normal patients at one site will have their primaquine treatment observed each day at the treatment centre by a qualified member of the staff designated by the principal investigator. Study patients will be observed for 60 minutes after drug administration for vomiting. Any patient who vomits during the first half-hour observation period will be retreated with the same dose of drug and observed for an additional 30 minutes. If the patient vomits in the second period they should receive half the drug. This will simply be noted and no further doses of primaquine given that day; doses will be given from the next day onwards as normal. A slightly extended case record form (CRF) will be used to record the timing of administration of primaquine doses in a tabular format.
5. Patients with G6PD deficiency discovered at baseline Patients judged to be G6PD deficient will receive counselling in terms of what the diagnosis means, how they should avoid certain drugs and to show the G6PD card every time they buy drugs from a pharmacy/drug store or visit their doctors. They will be provided with a G6PD deficiency card listing drugs they should avoid.
6. Follow-up Prior to going home on day 0, Patients will also be provided with clear verbal instructions in terms of self-monitoring for features of haemolysis, and advised to attend if any of these occur. All patients will be advised to return if they experience any side-effects. The Patient Information Sheet explains this and specifically refers to the symptom of dark urine.

   The patient will re-attend for follow-up at day 2, day 7 and day 14 and the following information recorded
   * Medical and medication history
   * Physical examination including vital signs
   * Capillary blood sample (finger prick)

     * Haemoglobin measurement
     * Dried blood spots (d7 and d14) for primaquine and carboxyprimaquine.
     * Day14 G6PD activity measured by the Biosensor (subset of patients)
   * Adverse events assessment focussing on patients who require hospitalisation
7. Haemolysis and stopping primaquine Based on the extensive work already undertaken on the G6PD RDT, and with appropriate care, primaquine-induced haemolysis should not be a significant problem in this study. However, it is important to stop primaquine in individuals with signs of haemolysis, whatever the result from the initial G6PD RDT.

Haemolysis is likely to manifest itself as early as first 48 hours after commencement of primaquine. The main symptoms are dark urine (macroscopic haemoglobinuria) and weakness / tiredness due to an acute fall in haemoglobin.

The following criteria will be used to define an episode of haemolysis that requires primaquine to be stopped (and not reintroduced):

* Either a drop in haemoglobin concentration by more than 2g/dl compared to baseline
* Or an absolute haemoglobin concentration of less than 7 g/dl at any time The healthcare worker may also stop primaquine administration for reasons outside these criteria. If necessary patients will be admitted for management, or referred / transferred elsewhere, as per local practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children >6 months
* Confirmed diagnosis of Plasmodium vivax mono-infection
* Ability to swallow oral medication
* Participant (or parent/guardian if <15 years old) is willing and able to give documented informed consent and comply with study requirements

Exclusion Criteria:

* Severe malaria (see World Health Organisation definition)
* P. falciparum infection
* Pregnancy or lactation
* Hypersensitivity (allergy) to primaquine or chloroquine
* Presence of any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study e.g. other acute febrile conditions or chronic disease
* Ongoing involvement in another research study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CareStart™ G6PD rapid test compared to a genotyping result as gold-standard | 3 years
Specificity of CareStart™ G6PD rapid test compared to a genotyping result as gold-standard | 3 years

SECONDARY OUTCOMES:
Percentage of P. vivax patients receiving a correct primaquine prescription after G6PD testing compared to using phenotype as gold standard | 3 years
Level of primaquine metabolite in dried blood spots collected after treatment | 2, 7 and 14 days
  Day 2, 7, 14
Level of whole blood carboxyprimaquine at day 7 | 7 days
Level of whole blood carboxyprimaquine at day 14 | 14 days
The degree to which healthcare workers act appropriately on the results of G6PD testing in terms of primaquine prescription | 3 years
Barriers to long-term use of the approach based on a qualitative questionnaire-based survey | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ghulam Rahim Awab MD, Jalalabad, Nangarha, Afghanistan

IPD SHARING:
Plan to Share IPD: No